CLINICAL TRIAL: NCT04445532
Title: Acquisition of Blood and Tumor Tissue Samples From Patients With Hepatobiliary Tumors
Brief Title: Hepatobiliary Tumors Tissue Samples Acquisition
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: OrigiMed (Industry); GeneCast Biotechnology Co., Ltd. (Industry); YuceBio Technology Co., Ltd. (Unknown); Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JS-2296
Record Dates: First submitted 2020-06-18; First posted 2020-06-24 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma; Gallbladder Cancer; Biliary Tract Cancer; Liver Cancer; Precancerous Condition; Benign Hepatobiliary Disease; Healthy, no Evidence of Disease
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Gallbladder Neoplasms; Biliary Tract Neoplasms; Liver Neoplasms; Precancerous Conditions | interventions — Gene Expression Profiling; Polymerase Chain Reaction; Mass Spectrometry; Immunohistochemistry; Methylation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, urine, feces, ascites, bile samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hepatobiliary tumor patients: benign or malignant hepatobiliary tumors patients
  Interventions: Other: Gene expression analysis; Other: Genomic analysis; Other: Protein expression analysis; Other: Proteomic profiling; Other: Polymerase chain reaction; Other: Mass spectrometry; Other: Immunohistochemistry; Other: Metabolomics profiling; Other: Methylation and epigenetic analysis; Other: Liquid biopsy analysis; Other: Laboratory biomarker analysis
- Benign Hepatobiliary Disease: chronic hepatitis, cirrhosis, and healthy control
  Interventions: Other: Gene expression analysis; Other: Genomic analysis; Other: Protein expression analysis; Other: Proteomic profiling; Other: Polymerase chain reaction; Other: Mass spectrometry; Other: Immunohistochemistry; Other: Metabolomics profiling; Other: Methylation and epigenetic analysis; Other: Liquid biopsy analysis; Other: Laboratory biomarker analysis

INTERVENTIONS:
Other: Gene expression analysis — Gene expression analysis
Other: Genomic analysis — Genomic analysis
Other: Protein expression analysis — Protein expression analysis
Other: Proteomic profiling — Proteomic profiling
Other: Polymerase chain reaction — Polymerase chain reaction
Other: Mass spectrometry — Mass spectrometry
Other: Immunohistochemistry — Immunohistochemistry
Other: Metabolomics profiling — Metabolomics profiling
Other: Methylation and epigenetic analysis — Methylation and epigenetic analysis
Other: Liquid biopsy analysis — Liquid biopsy analysis, such as cell-free DNA or circulating tumor cell analysis
Other: Laboratory biomarker analysis — Laboratory biomarker analysis (such as AFP, CA19-9, CEA)

SUMMARY:
Hepatobiliary tumors have a poor prognosis and high individual heterogeneity, so it is of great significance to find important prognostic markers and then screen out specific subgroups of people; meanwhile, chronic hepatitis, cirrhosis, and healthy control participants also need to show the evolution of tumors and discover specific diagnostic markers as a control group. Moreover, targeted therapy and immunotherapy make cancer treatment enter a new field, but only part of patients achieve response rates and reach clinical benefit. However, these drugs are expensive and can cause treatment-related adverse events. Therefore, reliable biomarkers identification is needed to help predict the response to these treatment options in order to screen patients with better responsiveness and avoid wasting money. Multi-omics research can reveal the characteristics of hepatobiliary tumors more deeply and find meaningful therapeutic targets.

Therefore, 450 patients at least 18 years of age with hepatobiliary tumors were included in this study.

DETAILED DESCRIPTION:
OBJECTIVES:

1. Observe the biomarkers of resectable hepatobiliary tumor recurrence (DFS) and survival (OS);
2. Observe the evolution of tumors and discover specific diagnostic markers as a control group.
3. Observe the response (ORR), progression (PFS) and survival (OS) biomarkers of targeted immunotherapy for advanced hepatobiliary tumors;
4. To elaborate on the multi-omics study of hepatobiliary tumors, to further subtype and find therapeutic targets

ELIGIBILITY:
Inclusion Criteria:

1. Be older than 18 years old;
2. ECOG 0-2 points;
3. May have received treatment;
4. Clinical consideration or diagnosis of benign and malignant hepatobiliary tumors; or chronic hepatitis, cirrhosis, or healthy control participants;
5. Patients may have received or are about to undergo surgery, chemotherapy, radiotherapy, targeted therapy, local therapy, immunotherapy, etc.;
6. Patients understand and are willing to sign written informed consent documents.

Exclusion Criteria:

1. The doctor thinks it is not suitable to enter the group (mental disorder or poor compliance, etc.)
2. Pregnant women;
3. Active or uncontrollable infections (fungi, bacteria, etc.);
4. Estimated survival time <12 weeks;
5. If the patient is receiving chronic anticoagulant therapy, the anticoagulant withdrawal should not be shorter than 3 days;
6. In the evaluation of the doctor, there is a risk of uncontrolled complications in the biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hepatobiliary cancer, benign hepatobiliary disease, and healthy Subjects will be recruited at Peking Union Medical College Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-10-11 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Collected samples | through study completion, an average of 5 years
  Collected normal tissue, tumor samples, blood, urine, feces, ascites, bile samples from patients with hepatobiliary cancers

SECONDARY OUTCOMES:
Biomarkers of resectable disease-free recurrence (DFS) and overall survival (OS) | through study completion, an average of 5 years
Biomarkers of evolution of tumors and discover specific diagnostic markers for hepatobiliary tumors | through study completion, an average of 5 years
Biomarkers of the efficacy of target and immunotherapy for advanced hepatobiliary tumors | through study completion, an average of 5 years
Multi-omics analysis to further type and find therapeutic targets | through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zhao, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Background] Banales JM, Cardinale V, Carpino G, Marzioni M, Andersen JB, Invernizzi P, Lind GE, Folseraas T, Forbes SJ, Fouassier L, Geier A, Calvisi DF, Mertens JC, Trauner M, Benedetti A, Maroni L, Vaquero J, Macias RI, Raggi C, Perugorria MJ, Gaudio E, Boberg KM, Marin JJ, Alvaro D. Expert consensus document: Cholangiocarcinoma: current knowledge and future perspectives consensus statement from the European Network for the Study of Cholangiocarcinoma (ENS-CCA). Nat Rev Gastroenterol Hepatol. 2016 May;13(5):261-80. doi: 10.1038/nrgastro.2016.51. Epub 2016 Apr 20. PMID 27095655
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Background] Zhou J, Sun HC, Wang Z, Cong WM, Wang JH, Zeng MS, Yang JM, Bie P, Liu LX, Wen TF, Han GH, Wang MQ, Liu RB, Lu LG, Ren ZG, Chen MS, Zeng ZC, Liang P, Liang CH, Chen M, Yan FH, Wang WP, Ji Y, Cheng WW, Dai CL, Jia WD, Li YM, Li YX, Liang J, Liu TS, Lv GY, Mao YL, Ren WX, Shi HC, Wang WT, Wang XY, Xing BC, Xu JM, Yang JY, Yang YF, Ye SL, Yin ZY, Zhang BH, Zhang SJ, Zhou WP, Zhu JY, Liu R, Shi YH, Xiao YS, Dai Z, Teng GJ, Cai JQ, Wang WL, Dong JH, Li Q, Shen F, Qin SK, Fan J. Guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2017 Edition). Liver Cancer. 2018 Sep;7(3):235-260. doi: 10.1159/000488035. Epub 2018 Jun 14. PMID 30319983
- [Background] Llovet JM, Montal R, Villanueva A. Randomized trials and endpoints in advanced HCC: Role of PFS as a surrogate of survival. J Hepatol. 2019 Jun;70(6):1262-1277. doi: 10.1016/j.jhep.2019.01.028. Epub 2019 Mar 31. PMID 30943423
- [Background] Valle JW, Borbath I, Khan SA, Huguet F, Gruenberger T, Arnold D; ESMO Guidelines Committee. Biliary cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2016 Sep;27(suppl 5):v28-v37. doi: 10.1093/annonc/mdw324. No abstract available. PMID 27664259
- [Background] Totoki Y, Tatsuno K, Covington KR, Ueda H, Creighton CJ, Kato M, Tsuji S, Donehower LA, Slagle BL, Nakamura H, Yamamoto S, Shinbrot E, Hama N, Lehmkuhl M, Hosoda F, Arai Y, Walker K, Dahdouli M, Gotoh K, Nagae G, Gingras MC, Muzny DM, Ojima H, Shimada K, Midorikawa Y, Goss JA, Cotton R, Hayashi A, Shibahara J, Ishikawa S, Guiteau J, Tanaka M, Urushidate T, Ohashi S, Okada N, Doddapaneni H, Wang M, Zhu Y, Dinh H, Okusaka T, Kokudo N, Kosuge T, Takayama T, Fukayama M, Gibbs RA, Wheeler DA, Aburatani H, Shibata T. Trans-ancestry mutational landscape of hepatocellular carcinoma genomes. Nat Genet. 2014 Dec;46(12):1267-73. doi: 10.1038/ng.3126. Epub 2014 Nov 2. PMID 25362482
- [Background] Cancer Genome Atlas Research Network. Electronic address: wheeler@bcm.edu; Cancer Genome Atlas Research Network. Comprehensive and Integrative Genomic Characterization of Hepatocellular Carcinoma. Cell. 2017 Jun 15;169(7):1327-1341.e23. doi: 10.1016/j.cell.2017.05.046. PMID 28622513
- [Background] Jiang Y, Sun A, Zhao Y, Ying W, Sun H, Yang X, Xing B, Sun W, Ren L, Hu B, Li C, Zhang L, Qin G, Zhang M, Chen N, Zhang M, Huang Y, Zhou J, Zhao Y, Liu M, Zhu X, Qiu Y, Sun Y, Huang C, Yan M, Wang M, Liu W, Tian F, Xu H, Zhou J, Wu Z, Shi T, Zhu W, Qin J, Xie L, Fan J, Qian X, He F; Chinese Human Proteome Project (CNHPP) Consortium. Proteomics identifies new therapeutic targets of early-stage hepatocellular carcinoma. Nature. 2019 Mar;567(7747):257-261. doi: 10.1038/s41586-019-0987-8. Epub 2019 Feb 27. PMID 30814741
- [Background] Zheng C, Zheng L, Yoo JK, Guo H, Zhang Y, Guo X, Kang B, Hu R, Huang JY, Zhang Q, Liu Z, Dong M, Hu X, Ouyang W, Peng J, Zhang Z. Landscape of Infiltrating T Cells in Liver Cancer Revealed by Single-Cell Sequencing. Cell. 2017 Jun 15;169(7):1342-1356.e16. doi: 10.1016/j.cell.2017.05.035. PMID 28622514
- [Background] Nakamura H, Arai Y, Totoki Y, Shirota T, Elzawahry A, Kato M, Hama N, Hosoda F, Urushidate T, Ohashi S, Hiraoka N, Ojima H, Shimada K, Okusaka T, Kosuge T, Miyagawa S, Shibata T. Genomic spectra of biliary tract cancer. Nat Genet. 2015 Sep;47(9):1003-10. doi: 10.1038/ng.3375. Epub 2015 Aug 10. PMID 26258846
- [Background] Sia D, Hoshida Y, Villanueva A, Roayaie S, Ferrer J, Tabak B, Peix J, Sole M, Tovar V, Alsinet C, Cornella H, Klotzle B, Fan JB, Cotsoglou C, Thung SN, Fuster J, Waxman S, Garcia-Valdecasas JC, Bruix J, Schwartz ME, Beroukhim R, Mazzaferro V, Llovet JM. Integrative molecular analysis of intrahepatic cholangiocarcinoma reveals 2 classes that have different outcomes. Gastroenterology. 2013 Apr;144(4):829-40. doi: 10.1053/j.gastro.2013.01.001. Epub 2013 Jan 4. PMID 23295441
- [Background] Villanueva A, Hoshida Y, Battiston C, Tovar V, Sia D, Alsinet C, Cornella H, Liberzon A, Kobayashi M, Kumada H, Thung SN, Bruix J, Newell P, April C, Fan JB, Roayaie S, Mazzaferro V, Schwartz ME, Llovet JM. Combining clinical, pathology, and gene expression data to predict recurrence of hepatocellular carcinoma. Gastroenterology. 2011 May;140(5):1501-12.e2. doi: 10.1053/j.gastro.2011.02.006. Epub 2011 Feb 12. PMID 21320499
- [Background] Toyoda H, Kumada T, Tada T, Niinomi T, Ito T, Kaneoka Y, Maeda A. Prognostic significance of a combination of pre- and post-treatment tumor markers for hepatocellular carcinoma curatively treated with hepatectomy. J Hepatol. 2012 Dec;57(6):1251-7. doi: 10.1016/j.jhep.2012.07.018. Epub 2012 Jul 20. PMID 22824818
- [Background] Wang Y, Li J, Xia Y, Gong R, Wang K, Yan Z, Wan X, Liu G, Wu D, Shi L, Lau W, Wu M, Shen F. Prognostic nomogram for intrahepatic cholangiocarcinoma after partial hepatectomy. J Clin Oncol. 2013 Mar 20;31(9):1188-95. doi: 10.1200/JCO.2012.41.5984. Epub 2013 Jan 28. PMID 23358969
- [Background] Bridgewater J, Lopes A, Wasan H, Malka D, Jensen L, Okusaka T, Knox J, Wagner D, Cunningham D, Shannon J, Goldstein D, Moehler M, Bekaii-Saab T, McNamara MG, Valle JW. Prognostic factors for progression-free and overall survival in advanced biliary tract cancer. Ann Oncol. 2016 Jan;27(1):134-40. doi: 10.1093/annonc/mdv483. Epub 2015 Oct 19. PMID 26483051
- [Background] Llovet JM, Montal R, Sia D, Finn RS. Molecular therapies and precision medicine for hepatocellular carcinoma. Nat Rev Clin Oncol. 2018 Oct;15(10):599-616. doi: 10.1038/s41571-018-0073-4. PMID 30061739
- [Background] Havel JJ, Chowell D, Chan TA. The evolving landscape of biomarkers for checkpoint inhibitor immunotherapy. Nat Rev Cancer. 2019 Mar;19(3):133-150. doi: 10.1038/s41568-019-0116-x. PMID 30755690
- [Background] Finn RS, Ryoo BY, Merle P, Kudo M, Bouattour M, Lim HY, Breder V, Edeline J, Chao Y, Ogasawara S, Yau T, Garrido M, Chan SL, Knox J, Daniele B, Ebbinghaus SW, Chen E, Siegel AB, Zhu AX, Cheng AL; KEYNOTE-240 investigators. Pembrolizumab As Second-Line Therapy in Patients With Advanced Hepatocellular Carcinoma in KEYNOTE-240: A Randomized, Double-Blind, Phase III Trial. J Clin Oncol. 2020 Jan 20;38(3):193-202. doi: 10.1200/JCO.19.01307. Epub 2019 Dec 2. PMID 31790344
- [Background] Taylor MH, Lee CH, Makker V, Rasco D, Dutcus CE, Wu J, Stepan DE, Shumaker RC, Motzer RJ. Phase IB/II Trial of Lenvatinib Plus Pembrolizumab in Patients With Advanced Renal Cell Carcinoma, Endometrial Cancer, and Other Selected Advanced Solid Tumors. J Clin Oncol. 2020 Apr 10;38(11):1154-1163. doi: 10.1200/JCO.19.01598. Epub 2020 Jan 21. PMID 31961766
- [Background] Sirica AE, Gores GJ, Groopman JD, Selaru FM, Strazzabosco M, Wei Wang X, Zhu AX. Intrahepatic Cholangiocarcinoma: Continuing Challenges and Translational Advances. Hepatology. 2019 Apr;69(4):1803-1815. doi: 10.1002/hep.30289. Epub 2019 Mar 25. PMID 30251463
- [Background] Flaherty KT, Gray R, Chen A, Li S, Patton D, Hamilton SR, Williams PM, Mitchell EP, Iafrate AJ, Sklar J, Harris LN, McShane LM, Rubinstein LV, Sims DJ, Routbort M, Coffey B, Fu T, Zwiebel JA, Little RF, Marinucci D, Catalano R, Magnan R, Kibbe W, Weil C, Tricoli JV, Alexander B, Kumar S, Schwartz GK, Meric-Bernstam F, Lih CJ, McCaskill-Stevens W, Caimi P, Takebe N, Datta V, Arteaga CL, Abrams JS, Comis R, O'Dwyer PJ, Conley BA; NCI-MATCH Team. The Molecular Analysis for Therapy Choice (NCI-MATCH) Trial: Lessons for Genomic Trial Design. J Natl Cancer Inst. 2020 Oct 1;112(10):1021-1029. doi: 10.1093/jnci/djz245. PMID 31922567
- [Background] Nault JC, Villanueva A. Biomarkers for Hepatobiliary Cancers. Hepatology. 2021 Jan;73 Suppl 1:115-127. doi: 10.1002/hep.31175. Epub 2020 Nov 29. PMID 32045030